CLINICAL TRIAL: NCT04409366
Title: One- Versus Two-Stage Aesthetic Crown Lengthening for Restorative Purposes: A Randomized Controlled Trial.
Brief Title: One- Versus Two-Stage Aesthetic Crown Lengthening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Crown Lengthening RCT
Record Dates: First submitted 2020-05-26; First posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Patients in Need of Surgical CL in the Anterior Maxillary Sextant for Restorative Purposes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Crown Lengthening; CCL (Active Comparator): Using the surgical guide, submarginal internal bevel incisions were performed on the buccal aspect of the affected teeth. A full-thickness flap was raised up to the mucogingival junction (Dominguez et al., 2020). Ostectomy and osteoplasty were carried out by means of rotatory instruments and surgical chisels, as necessary, to achieve the necessary space between the bone crest and the restorative margin according to the presurgical plan. The CEJ was not the reference point since, in many cases, the position of the final margin of the restoration was planned apical to the actual position of the CEJ. Exposed root surfaces were carefully instrumented manually with curettes and, finally, vertical internal mattress sutures were placed to position the gingival margin at the level of the margin of the planned restoration. Sutures were removed after 7 days.
  Interventions: Other: Conventional Crown Lengthening (CCL)
- Two-stage Crown Lengthening (SCL) (Experimental): In the first surgical intervention, intrasulcular incisions were performed and a full thickness flap was raised up to the mucogingival junction. Ostectomy and osteoplasty were performed to establish the space for supracrestal tissue attachment, following the restorative plan and using the presurgical blueprint as the reference to determine the final position of the restoration margin, instead of the CEJ (Lee, 2004). Then the flaps were repositioned and secured with internal mattress sutures, placing the gingival margin at the original level. Sutures were removed at 7 days. In the second stage, after 3-4 months, minor gingival recontouring was performed, if necessary, to attain the desired gingival margin position according to the presurgical plan
  Interventions: Other: Two-stage Crown Lengthening (SCL)

INTERVENTIONS:
Other: Conventional Crown Lengthening (CCL) — Using the surgical guide, submarginal internal bevel incisions were performed on the buccal aspect of the affected teeth. A full-thickness flap was raised up to the mucogingival junction (Dominguez et al., 2020). Ostectomy and osteoplasty were carried out by means of rotatory instruments and surgical chisels, as necessary, to achieve the necessary space between the bone crest and the restorative margin according to the presurgical plan. The CEJ was not the reference point since, in many cases, the position of the final margin of the restoration was planned apical to the actual position of the CEJ. Exposed root surfaces were carefully instrumented manually with curettes and, finally, vertical internal mattress sutures were placed to position the gingival margin at the level of the margin of the planned restoration. Sutures were removed after 7 days
  Arms: Conventional Crown Lengthening; CCL
Other: Two-stage Crown Lengthening (SCL) — In the first surgical intervention, intrasulcular incisions were performed and a full thickness flap was raised up to the mucogingival junction. Ostectomy and osteoplasty were performed to establish the space for supracrestal tissue attachment, following the restorative plan and using the presurgical blueprint as the reference to determine the final position of the restoration margin, instead of the CEJ (Lee, 2004). Then the flaps were repositioned and secured with internal mattress sutures, placing the gingival margin at the original level. Sutures were removed at 7 days. In the second stage, after 3-4 months, minor gingival recontouring was performed, if necessary, to attain the desired gingival margin position according to the presurgical plan.
  Arms: Two-stage Crown Lengthening (SCL)

SUMMARY:
This randomized controlled trial was aimed at assessing the efficacy of a two-stage crown lengthening intervention (SCL) for restorative purposes in the aesthetic zone compared with a one-stage crown lengthening procedure (CCL).

DETAILED DESCRIPTION:
Subjects were randomly allocated to receive SCL or CCL. SCL consisted of full thickness flaps followed by bone recontouring and minor gingivectomy 4 months postoperatively, if required. In CCL, osseous recontouring after sub-marginal incisions was performed, followed by flap repositioning. Records were obtained at baseline, 4 months (only in SCL), 6 and 12 months. Primary outcome was the precision in achieving a predetermined gingival margin position. Other outcomes were changes in the gingival margin position and keratinized tissue width (KTW) at 12 months, and patient-reported outcomes (PROMs) using the OHIP-14 tool.

ELIGIBILITY:
Inclusion Criteria:

* older than eighteen years of age;
* more than 20 teeth in the mouth;
* with full mouth plaque and bleeding scores lower than 15%; and
* without probing pocket depth and/or attachment loss >4 mm

Exclusion Criteria:

* Pregnant women or breastfeeding
* smokers
* treated with antimicrobial and/or anti-inflammatory drugs within two months prior to entering the study
* currently undergoing orthodontic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
T1-T4 | Baseline-12 months
  The difference in mm between the ideal gingival margin (T1) and the position of the gingival margin at 12 months (T4).

SECONDARY OUTCOMES:
Clinical Crown Length | At baseline, 6- and 12-month
  Distance from the gingival margin to the incisal edge on the midbuccal.Measured in mm.
Amount of keratinized tissue | At baseline, 6- and 12-month
  Distance from the gingival margin to the mucogingival junction on the midbuccal.Measured in mm.
Gingival display upon smiling | At baseline, 6- and 12-month
  Distance from the gingival margin of the central incisors to the lower edge of the upper lip. Measured in mm.
Supracrestal tissue dimension | At baseline, 6- and 12-month
  Distance from the gingival margin to the alveolar bone crest (GM-ABC) as determined by bone sounding following local anesthesia. Measured in mm.

REFERENCES:
- [Derived] Gonzalez-Martin O, Carbajo G, Rodrigo M, Montero E, Sanz M. One- versus two-stage crown lengthening surgical procedure for aesthetic restorative purposes: A randomized controlled trial. J Clin Periodontol. 2020 Dec;47(12):1511-1521. doi: 10.1111/jcpe.13375. Epub 2020 Oct 20. PMID 32997836